CLINICAL TRIAL: NCT04616586
Title: A Study Comparing the Efficacy and Safety of Standard of Care With or Without Siltuximab in Selected Hospitalized Patients With Viral Acute Respiratory Distress Syndrome (SILVAR)
Brief Title: SILtuximab in Viral ARds (SILVAR) Study
Acronym: SILVAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The REMAP-CAP and RECOVERY substudy results appear to support the survival benefit of tocilizumab in corticosteroid-treated or untreated patients with critically ill COVID-19-associated ARDS.
Sponsor: RECORDATI GROUP (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EUSA SYL 0004
Record Dates: First submitted 2020-10-10; First posted 2020-11-05 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-01

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Diseases; Pneumonia; Respiratory Tract Infections; Respiratory Tract Disease
Keywords: Siltuximab; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases; Pneumonia; Respiratory Tract Infections; Respiratory Tract Diseases | interventions — siltuximab; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized (2:1), double-blind, parallel-arm, placebo-controlled, Phase 3 clinical trial of 1-3 doses of siltuximab 11 mg/kg IV over 1 hour plus SOC vs. matched-volume normal saline (NS) IV over 1 hour plus SOC in 555 patients with SARS-CoV-2 previously treated with corticosteroids or another respiratory virus infection with elevated CRP levels who have developed serious respiratory complications
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At all times, randomized study treatment assignment information will be kept confidential and will not be released to the patient, investigator, the study staff (except the pharmacist), or the Sponsor's Study Team until following the conclusion of the study, except as described below.
  At the initiation of the study, the study site will be instructed on procedures for breaking the blind. Blinding codes should be broken only in emergency situations for reasons of patient safety. If a patient has an AE that may be considered treatment-related, treatment for the AE should be administered as if the patient is receiving siltuximab. Whenever possible, the investigator should contact the Sponsor's Medical Monitor before breaking the blind. When the blind for a patient has been broken, the reason must be fully documented. The patient for whom the blind has been broken will not receive further doses of study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Drug - Siltuximab
  Interventions: Drug: Siltuximab
- Arm B (Other): Comparator - Normal Saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Siltuximab — 11 mg/kg IV administered over 1 hour
  Other Names: Sylvant
  Arms: Arm A
Other: Normal Saline — IV administered over 1 hour
  Arms: Arm B

SUMMARY:
This study will evaluate the efficacy and safety of siltuximab compared with normal saline in combination with standard of care (SOC) in selected hospitalized patients with COVID-19 previously treated with corticosteroids or another respiratory virus infection associated with acute respiratory distress syndrome (ARDS) and elevated C-reactive protein (CRP) levels.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized (2:1), double-blind, parallel-arm, placebo-controlled, Phase 3 clinical trial of 1-3 doses of siltuximab 11 mg/kg IV over 1 hour plus SOC vs. matched-volume normal saline (NS) IV over 1 hour plus SOC in 555 patients with SARS CoV-2 previously treated with corticosteroids or another respiratory virus infection with elevated CRP levels who have developed serious respiratory complications.

The randomization will be stratified by age (<65, ≥65 years), respiratory virus infection (confirmed SARS-CoV-2, other), and MIV status (yes, no). Crossover between treatment arms will not be allowed.

All patients will receive ARDS SOC following the official American Thoracic Society/European Society of Intensive Care Medicine/Society of Critical Care Medicine clinical practice guideline13 and/or the World Health Organization's (WHO's) clinical management of severe acute respiratory infection when COVID-19 disease is suspected (WHO Interim Guidance 202014 or other local guidance). Patients may continue receiving their corticosteroid (up to a cumulative maximum dexamethasone or equivalent dose of 60 mg [except to treat treatment-emergent reactions or comorbid conditions]) or antiviral therapy (except aminoquinoline compounds and convalescent plasma) at the same or lower doses if started at least 4 days (corticosteroid therapy) or at least 2 days (antiviral therapy) prior to randomization. Patients randomized to Arm A will additionally receive siltuximab 11 mg/kg IV administered over 1 hour, while patients randomized to Arm B will additionally receive IV NS administered over 1 hour, with opportunity to repeat their assigned study treatment once or twice at least 2 days apart on or after Day 3 as their clinical condition and/or laboratory testing dictate.

ELIGIBILITY:
Inclusion Criteria:

* Positive microbiological evidence of SARS-CoV-2 or another respiratory virus infection (eg, other coronaviruses, respiratory syncytial virus, influenza virus) following institutional diagnostic standards
* Clinical and radiological diagnosis of pulmonary infection requiring noninvasive or mechanical invasive ventilatory support plus administration of rising supplemental oxygen concentrations
* Treatment of SARS-CoV-2-infected patients with dexamethasone (or equivalent) administered by mouth or intravenous (IV) injection
* Diagnosis of ARDS (PaO2/FiO2 ≤200 with positive end-expiratory pressure ≥5 cmH2O) in accordance with Berlin 2012 criteria1 (measured on or after the fourth day after the start of corticosteroid therapy in those patients for whom it was prescribed)
* Serum CRP level greater than upper limit of normal (measured on or after the third day after the start of corticosteroid therapy in those patients for whom it was prescribed) on 2 consecutive days
* Age ≥12 years

Exclusion Criteria:

* Active bacterial or fungal infection, human immunodeficiency virus (HIV), HHV, Epstein-Barr virus, or other non-respiratory virus infection, or tuberculosis requiring initiation of anti-infective therapy
* Prior treatment with an agent targeting the IL-6 signaling pathway
* Current treatment in another therapeutic clinical trial (other than expanded remdesivir access protocol)
* Start of new immunosuppressive therapy (including but not limited to corticosteroids and cytokine signaling pathway inhibitors) within 4 days prior to study entry (randomization); start of new antiviral treatment (including but not limited to nucleoside analogues, aminoquinoline compounds, and convalescent plasma) within 2 days prior to randomization; or received a live vaccine at any time prior to randomization, or plan to receive a live vaccine during the study

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality | Day 28
  28-day all-cause mortality

SECONDARY OUTCOMES:
Time to 7-category ordinal scale of clinical status improvement (T7COSCSI) | Up to 60 days
  Time to 7-category ordinal scale of clinical status improvement (T7COSCSI)
Ventilator-free days (VFDs) within 28 days | Up to 28 days
  Ventilator-free days (VFDs) within 28 days
Organ failure-free days (OFFD) | Up to 60 days
  Organ failure-free days (OFFD)
Intensive care unit length of stay (ICU LOS) | Up to 60 days
  Intensive care unit length of stay (ICU LOS)
Hospital length of stay (HLOS) | Up to 60 days
  Hospital length of stay (HLOS)
In-hospital all-cause mortality (IHACM) | Up to 60 days
  In-hospital all-cause mortality (IHACM)
60-day all-cause mortality (60DACM) | Up to 60 days
  60-day all-cause mortality (60DACM)
Time to oxygenation improvement (TOI) | Up to 60 days
  Time to oxygenation improvement (TOI)
Duration of supplemental oxygen (DSO) | Up to 60 days
  Duration of supplemental oxygen (DSO)
Chest radiographic improvement (CRI) | Up to 60 days
  Chest radiographic improvement (CRI)
Time to National Early Warning Score 2 improvement (TNEWS2I) | Up to 60 days
  Time to National Early Warning Score 2 improvement (TNEWS2I)
Treatment-emergent adverse events (TEAEs) | Up to 60 days
  Treatment-emergent adverse events (TEAEs)
Plasma siltuximab concentrations (PSCs) | Up to 60 days
  Plasma siltuximab concentrations (PSCs)
Anti-siltuximab antibodies (ASA) | Up to 60 days
  Anti-siltuximab antibodies (ASA)

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Shahid, MD, Ph.D, Principal Investigator — Participating Site
Locations (2):
- United States (2):
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Atrium Health, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No